CLINICAL TRIAL: NCT05659992
Title: Single Arm,open Label,phase I Clinical Study of Venetoclax Combined with CACAG Regimen in the Treatment of Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Clinical Study of Venetoclax Combined with CACAG Regimen in the Treatment of Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, doctor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2022-240
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Venetoclax; CACAG; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): Experimental: Venetoclax combined CACAG regimen for newly diagnosed AML. All recipients in this arm received azacytidine, cytarabine.aclamycin, chidamide,venetoclax and granulocyte colony-stimulating factor.Azacytidine was uesd as 75 mg/m2/day from day-1 to day-7.Cytarabine was uesd as 75 mg/m2 bid from day-1 to day-5. Aclamycin was uesd as 10 mg/m2/day on day1,3,5). Chidamide was uesd as 30 mg/day twice per week for 2 weeks. Venetoclax was uesd as 100 mg on day 1, 200 mg on day 2, 400mg from day-3 to day-14.Granulocyte colony-stimulating factor was uesd as 5ug/kg/day from day 0 until agranulocytosis recovery.
  Interventions: Drug: azacytidine;cytarabine;aclamycin;Chidamide;venetoclax;granulocyte

INTERVENTIONS:
Drug: azacytidine;cytarabine;aclamycin;Chidamide;venetoclax;granulocyte — 1. azacytidine (75 mg/m2/day, days 1 to 7).
  2. cytarabine (75 mg/m2 bid, days 1 to 5).
  3. aclamycin (10 mg/m2/day, day1,3,5).
  4. Chidamide (30 mg/day , days 0,3).
  5. venetoclax (100 mg day 1, 200 mg day 2, 400mg days 3 to 14 ).
  6. granulocyte colony-stimulating factor (5ug/kg/day, day 0 until agranulocytosis recovery)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of venetoclax combined with CACAG regimen in the treatment of newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
Despite the availability of hematopoietic stem cell transplantation and the emergence of many new therapeutic drugs, the prognosis of newly diagnosed acute myeloid leukemia is still poor. In order to improve the outcome of patients with de novo AML, participants developed a venetoclax combined with CACAG regimen in the treatment of de novo AML. In this study, participants intent to evaluate the efficacy and safety of venetoclax combined with CACAG regimen in the treatment of newly diagnosed AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to understand and willing to sign the informed consent form (ICF).
* All patients should aged 14 to75 years,no gender limitation.
* Patients who are newly diagnosed with AML.
* Liver function: ALT and AST≤2.5 times the upper limit of normal ,bilirubin≤2 times the upper limit of normal;
* Renal function: creatinine ≤the upper limit of normal;
* Patients without any uncontrolled infections , without organ dysfunction or without severe mental illness;
* The score of Eastern Cooperative Oncology Group (ECOG) is 0-3,and the predicted survival ≥ 4 months.
* Patients without severe allergic constitution.

Exclusion Criteria:

* Patients with allergy or contraindication to the study drug;
* Female patients who are pregnant or breast-feeding.
* Patients with active infection
* Patients with a known history of alcohol or drug addiction on the basis that there could be a higher risk of non-compliance to study treatment;
* Patients with mental illness or other states unable to comply with the protocol;
* Less than 6 weeks after surgical operation of important organs.
* Liver function: ALT and AST>2.5 times the upper limit of normal ,bilirubin>2 times the upper limit of normal;Renal function: creatinine >the upper limit of normal;
* The patient is not suitable for this clinical trial (poor compliance, substance abuse, etc.)

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 month after study treatment
  Defined as the percentage of participants achieving a best overall response of complete response (CR), CR with incomplete blood count recovery (CRi), or partial response (PR).

SECONDARY OUTCOMES:
Rate of Minimal Residual Disease (MRD)-Negative Response: | after two courses of chemotherapy (each course is 28 days)
  Percentage of participants who achieved MRD-negative response, defined as < 1 leukemia cell per 10,000 leukocytes as assessed by flow cytometry or < 0.01% as assessed by PCR of a bone marrow aspirate.
Progression Free Survival (PFS) | 180 days after study treatment
  PFS was defined as time from the date joining the clinical study to the date of disease progression (PD) or date of death due to any cause, whichever occurred first.
Overall Survival (OS) | 180 days after study treatment
  Defined as the time from joining the clinical study to death due to any cause.
Rate of Participants With Adverse Events | Through 28 days post last study medication administration
  Percentage of Participants with 3 or 4 grade Adverse Events reported through 28 days post last study medication administration.
Partial Remission (PR) Rate: | 1 month after study treatment
  All hematologic criteria of CR; decrease of bone marrow blast percentage to 5 to 25 percent; and decrease of pre-treatment bone marrow blast percentage by at least 50 percent.
Complete Remission (CR) Rate | 1 month after study treatment
  Defined in accordance with the IWG Response Criteria in AML. Bone marrow blasts <5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions.
CR with Incomplete Blood Count Recovery Rate | 1 month after study treatment
  All CR criteria except for residual neutropenia (<1.0 x 109/L (1000/µL)) or thrombocytopenia (<100 x 109/L (100,000/µL)

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu Liu, doctor, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Q, Yang J, Lv L, Zhang X, Li M, Xu L, Huang S, Jing Y, Dou L. Phase 2 study of chidamide in combination with CAG and venetoclax-azacitidine in older patients with newly diagnosed acute myeloid leukemia. Front Immunol. 2025 Feb 26;16:1525110. doi: 10.3389/fimmu.2025.1525110. eCollection 2025. PMID 40079007